CLINICAL TRIAL: NCT04638101
Title: Building the Path to Resilience in Preterm Infants: a Neuroimaging Investigation of the Impact of Multisensory and Neurocognitive Interventions Concern: Mindfulness-based Intervention
Brief Title: Building the Path to Resilience in Preterm Infants: Mindfulness-based Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Principal Investigator, Petra Hüppi, Professor, Pediatric Clinical Research Platform
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-00175
Record Dates: First submitted 2020-10-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Preterm Birth; Cognitive Dysfunction; Behavioral Problem
MeSH Terms: conditions — Premature Birth; Cognitive Dysfunction; Problem Behavior

STUDY DESIGN:
Intervention Model Description: For young adolescents enrolled in the randomised controlled trial design, families were randomised either to the intervention group or the waiting group.
  Participants enrolled in the RCT completed three assessments at three different time points: Time 1, Time 2, Time 3. Participants from the intervention group participated in Mindfulness-based intervention between Time 1 and Time 2. Participants from the waiting group took part in the Mindfulness-based intervention between Time 2 and Time 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (RCT) (Experimental): Participants from the intervention group participated in the mindfulness-based intervention between Time 1 and Time 2.
  Interventions: Behavioral: Mindfulness-based intervention
- Waiting group (RCT) (Experimental): Participants from the waiting group took part in the mindfulness-based intervention between Time 2 and Time 3.
  Interventions: Behavioral: Mindfulness-based intervention

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — Mindfulness-based intervention: The proposed MBI was designed based on well-known MBI programs including Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy and adapted to adolescents' needs and language. The program consisted of 8 weekly sessions in groups of up to 8 participants, lasting 1h30. Two MBI groups were offered per week (Wednesdays and Fridays) and participants had the possibility to choose the most convenient day for them. Two instructors were present for each group throughout the intervention.For each session one theme was addressed, such as attention and the stabilisation of the focus of attention, bodily sensations, breath, emotions, thoughts, compassion, stress, stress reactivity and coping strategies.

SUMMARY:
Yearly 15 million babies worldwide are born too soon. 10% of these preterm births occur very early before 32 weeks of gestation and these newborns are at high risk for neurodevelopmental disorders later in life. Neurocognitive disorders now touch 27% of the European population, and 5% or 3.3 million children suffer from social and learning difficulties, including attention-deficit hyperactivity disorders and autism, whose rates are increasing and prematurity contributes to this rise. Cognition, and socio-emotional competence are based on intact brain structure and functions that are formed early in development, both pre- and post-natally, and are heavily influenced by environment. Ramon y Cajal in his studies on the making of the brain clearly stated: "The total arborisation of a neuron represents the graphic history of conflicts suffered during its developmental life". Understanding how environment affects early brain development and defining timing and mode of early interventions to enhance brain development in high risk populations, such as preterm infants, is currently acknowledged as a fundamental endeavor for the scientific community (see guidelines of the National Scientific Council for the Developing Child). Interventions to improve and maintain cognitive and socio-emotional skills are to become an essential tool of medical care for high-risk infants. The goal of this study is to test the impact of a Mindfulness-based intervention - considered to target brain networks previously described as affected by prematurity and improve socio-emotional and executive functions. Mindfulness based intervention (intentional self-regulation of attention) will be performed in 10-13 year old preterm children, both from our prior studied preterm cohorts. Overall, our planned research will fill an important gap in our theoretical understanding of the brain vulnerability linked to prematurity. Even more importantly, the compelling issue of how to build cognitive and emotional resilience in preterm children will be addressed by preventing the onset of difficulties and reducing them with appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

* born before 32 gestational weeks

Exclusion Criteria:

* severe sensory or physical disabilities (cerebral palsy, blindness, hearing loss)
* intelligence quotient below 70
* not French speaking

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Behaviour Rating Inventory of Executive Function, parent questionnaire (BRIEF; Gioia, Isquith, Guy, and Kenworthy (2000)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  Executive competences of young adolescents were assessed using the Behaviour Rating Inventory of Executive Function - parent questionnaire version (BRIEF) evaluating attention, hyperactivity and impulsivity in everyday life. The BRIEF comprises 86 items over two standardised subscales, the Behavioural Regulation Index (BRI) and the Metacognition Index (MI), as well as a global score called the Global Executive Composite (GEC). These 3 scores will be used as a measure of executive function in daily life. Higher scores mean worse outcomes.
Behaviour Rating Inventory of Executive Function, parent questionnaire (BRIEF; Gioia, Isquith, Guy, and Kenworthy (2000)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  Executive competences of young adolescents were assessed using the Behaviour Rating Inventory of Executive Function - parent questionnaire version (BRIEF) evaluating attention, hyperactivity and impulsivity in everyday life. The BRIEF comprises 86 items over two standardised subscales, the Behavioural Regulation Index (BRI) and the Metacognition Index (MI), as well as a global score called the Global Executive Composite (GEC). These 3 scores will be used as a measure of executive function in daily life. Higher scores mean worse outcomes.
Behaviour Rating Inventory of Executive Function, parent questionnaire (BRIEF; Gioia, Isquith, Guy, and Kenworthy (2000)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  Executive competences of young adolescents were assessed using the Behaviour Rating Inventory of Executive Function - parent questionnaire version (BRIEF) evaluating attention, hyperactivity and impulsivity in everyday life. The BRIEF comprises 86 items over two standardised subscales, the Behavioural Regulation Index (BRI) and the Metacognition Index (MI), as well as a global score called the Global Executive Composite (GEC). These 3 scores will be used as a measure of executive function in daily life. Higher scores mean worse outcomes.
Strength and Difficulties Questionnaire, parent questionnaire (SDQ; Goodman (2001)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The SDQ parent questionnaire assess overall behaviour problems, emotional symptoms, hyperactivity and inattention, peer relationship problems, and prosocial behaviour. It rates participant's behaviour over the previous 6 months. The SDQ is scored on a Likert scale and includes 25 items, providing a Total Difficulties score. The Total Difficulties score will be use as a score of behavioural functionning in daily life. Higher scores mean worse outcomes.
Strength and Difficulties Questionnaire, parent questionnaire (SDQ; Goodman (2001)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The SDQ parent questionnaire assess overall behaviour problems, emotional symptoms, hyperactivity and inattention, peer relationship problems, and prosocial behaviour. It rates participant's behaviour over the previous 6 months. The SDQ is scored on a Likert scale and includes 25 items, providing a Total Difficulties score. The Total Difficulties score will be use as a score of behavioural functionning in daily life. Higher scores mean worse outcomes.
Strength and Difficulties Questionnaire, parent questionnaire (SDQ; Goodman (2001)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The SDQ parent questionnaire assess overall behaviour problems, emotional symptoms, hyperactivity and inattention, peer relationship problems, and prosocial behaviour. It rates participant's behaviour over the previous 6 months. The SDQ is scored on a Likert scale and includes 25 items, providing a Total Difficulties score. The Total Difficulties score will be use as a score of behavioural functionning in daily life. Higher scores mean worse outcomes.
KIDSCREEN-27 - Self-reported questionnaire (Robitail et al., 2007) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The KIDSCREEN-27 is a self-reported questionnaire providing an index of health-related quality of life in children and adolescents. This instrument scored on a Likert scale and includes 27 items, providing a total score. The total score will be used as a measure of quality of life. Higher scores mean better outcomes.
KIDSCREEN-27 - Self-reported questionnaire (Robitail et al., 2007) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The KIDSCREEN-27 is a self-reported questionnaire providing an index of health-related quality of life in children and adolescents. This instrument scored on a Likert scale and includes 27 items, providing a total score. The total score will be used as a measure of quality of life. Higher scores mean better outcomes.
KIDSCREEN-27 - Self-reported questionnaire (Robitail et al., 2007) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The KIDSCREEN-27 is a self-reported questionnaire providing an index of health-related quality of life in children and adolescents. This instrument scored on a Likert scale and includes 27 items, providing a total score. The total score will be used as a measure of quality of life. Higher scores mean better outcomes.
Social Goal Scale - Self-reported questionnaire (SGS; Patrick, Hicks, and Ryan (1997)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The SGS is a self-reported questionnaire providing an index of social responsiveness and of goals setting which ultimately gets you involve with some social work. This instrument scored on a Likert scale and includes 11 items providing one total score that will be used as a measure of social goal. Higher scores mean better outcomes.
Social Goal Scale - Self-reported questionnaire (SGS; Patrick, Hicks, and Ryan (1997)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The SGS is a self-reported questionnaire providing an index of social responsiveness and of goals setting which ultimately gets you involve with some social work. This instrument scored on a Likert scale and includes 11 items providing one total score that will be used as a measure of social goal. Higher scores mean better outcomes.
Social Goal Scale - Self-reported questionnaire (SGS; Patrick, Hicks, and Ryan (1997)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The SGS is a self-reported questionnaire providing an index of social responsiveness and of goals setting which ultimately gets you involve with some social work. This instrument scored on a Likert scale and includes 11 items providing one total score that will be used as a measure of social goal. Higher scores mean better outcomes.
Self-Compassion Scale - Short form - Self-reported questionnaire (SCS; Raes, Pommier, Neff, and Van Gucht (2011)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The SCS is a self-reported questionnaire comprising 12 items, which produces a total global score. The total global score will be used as a measure of self compassion. Higher scores mean better outcomes.
Self-Compassion Scale - Short form - Self-reported questionnaire (SCS; Raes, Pommier, Neff, and Van Gucht (2011)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The SCS is a self-reported questionnaire comprising 12 items, which produces a total global score. The total global score will be used as a measure of self compassion. Higher scores mean better outcomes.
Self-Compassion Scale - Short form - Self-reported questionnaire (SCS; Raes, Pommier, Neff, and Van Gucht (2011)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The SCS is a self-reported questionnaire comprising 12 items, which produces a total global score. The total global score will be used as a measure of self compassion. Higher scores mean better outcomes.
Letter-Number Sequencing (WISC-IV; Wechsler (2003)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The letter-number sequencing is a working memory task. Sequences of number and letters are read to the participant, and he/she is then asked to re-sequence the numbers in numerical order from lowest to highest and then to sequence the letters in alphabetical order. Standardised total scores will be used as a measure of working memory. Higher scores mean better outcomes.
Letter-Number Sequencing (WISC-IV; Wechsler (2003)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The letter-number sequencing is a working memory task. Sequences of number and letters are read to the participant, and he/she is then asked to re-sequence the numbers in numerical order from lowest to highest and then to sequence the letters in alphabetical order. Standardised total scores will be used as a measure of working memory. Higher scores mean better outcomes.
Letter-Number Sequencing (WISC-IV; Wechsler (2003)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The letter-number sequencing is a working memory task. Sequences of number and letters are read to the participant, and he/she is then asked to re-sequence the numbers in numerical order from lowest to highest and then to sequence the letters in alphabetical order. Standardised total scores will be used as a measure of working memory. Higher scores mean better outcomes.
Tempo Test Rekenen (De Vos, 1992) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The Tempo Test Rekenen is an arithmetic test consisting of 200 arithmetic number fact problems presented in five rows (one row with addition, one row with subtraction, one row with division, one row with multiplication, and one mixed problem row). Within each row, the problems increase in difficulty. Participant are asked to solve as many items as possible within 1 min per row. The total raw score will be age-adjusted for each participant and used as a measure of arithmetic competences. Higher scores mean better outcomes.
Tempo Test Rekenen (De Vos, 1992) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The Tempo Test Rekenen is an arithmetic test consisting of 200 arithmetic number fact problems presented in five rows (one row with addition, one row with subtraction, one row with division, one row with multiplication, and one mixed problem row). Within each row, the problems increase in difficulty. Participant are asked to solve as many items as possible within 1 min per row. The total raw score will be age-adjusted for each participant and used as a measure of arithmetic competences. Higher scores mean better outcomes.
Tempo Test Rekenen (De Vos, 1992) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The Tempo Test Rekenen is an arithmetic test consisting of 200 arithmetic number fact problems presented in five rows (one row with addition, one row with subtraction, one row with division, one row with multiplication, and one mixed problem row). Within each row, the problems increase in difficulty. Participant are asked to solve as many items as possible within 1 min per row. The total raw score will be age-adjusted for each participant and used as a measure of arithmetic competences. Higher scores mean better outcomes.
Affect Recognition (NEPSY-II; Korkman, Kirk, and Kemp (2007) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The affect recognition subtest assesses the ability to recognise facial emotional expressions (happy, sad, anger, fear, disgust, and neutral) from photographs of children's faces in several matching tasks. In the first task, the participant selected one of the four faces that depicted the same emotion as a child's face at the top of the page. In a second task, the participant selected two photographs of faces that displayed the same affect from a selection of four photographs. Finally, the participant examined a photograph of a child's face for 5 seconds, and then from memory, selected two photographs that matched the same emotion as the face previously shown. Standardised scores will be used. Higher scores mean better outcomes.
Affect Recognition (NEPSY-II; Korkman, Kirk, and Kemp (2007) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The affect recognition subtest assesses the ability to recognise facial emotional expressions (happy, sad, anger, fear, disgust, and neutral) from photographs of children's faces in several matching tasks. In the first task, the participant selected one of the four faces that depicted the same emotion as a child's face at the top of the page. In a second task, the participant selected two photographs of faces that displayed the same affect from a selection of four photographs. Finally, the participant examined a photograph of a child's face for 5 seconds, and then from memory, selected two photographs that matched the same emotion as the face previously shown. Standardised scores will be used. Higher scores mean better outcomes.
Affect Recognition (NEPSY-II; Korkman, Kirk, and Kemp (2007) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The affect recognition subtest assesses the ability to recognise facial emotional expressions (happy, sad, anger, fear, disgust, and neutral) from photographs of children's faces in several matching tasks. In the first task, the participant selected one of the four faces that depicted the same emotion as a child's face at the top of the page. In a second task, the participant selected two photographs of faces that displayed the same affect from a selection of four photographs. Finally, the participant examined a photograph of a child's face for 5 seconds, and then from memory, selected two photographs that matched the same emotion as the face previously shown. Standardised scores will be used. Higher scores mean better outcomes.
Theory of Mind (NEPSY-II; Korkman et al. (2007)) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The theory of mind subtest measures understanding of mental functions and other people's perspectives.
  In the first task, questions are asked to the participant about different verbal scenarios measuring understanding of beliefs, intentions, others' thoughts, ideas and comprehension of figurative language. In the second task, participants have to match facial emotional expressions, from photographs of children's faces, to a scenario. The total raw score willl be age-adjusted. Higher scores mean better outcomes.
Theory of Mind (NEPSY-II; Korkman et al. (2007)) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The theory of mind subtest measures understanding of mental functions and other people's perspectives.
  In the first task, questions are asked to the participant about different verbal scenarios measuring understanding of beliefs, intentions, others' thoughts, ideas and comprehension of figurative language. In the second task, participants have to match facial emotional expressions, from photographs of children's faces, to a scenario. The total raw score willl be age-adjusted. Higher scores mean better outcomes.
Theory of Mind (NEPSY-II; Korkman et al. (2007)) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The theory of mind subtest measures understanding of mental functions and other people's perspectives.
  In the first task, questions are asked to the participant about different verbal scenarios measuring understanding of beliefs, intentions, others' thoughts, ideas and comprehension of figurative language. In the second task, participants have to match facial emotional expressions, from photographs of children's faces, to a scenario. The total raw score willl be age-adjusted. Higher scores mean better outcomes.
Flanker Visual Filtering Task (Christ, Kester, Bodner, & Miles, 2011) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The Flanker Visual Filtering Task was used to assess attentional control and information processing speed. Each trial showed a horizontal row of five fish. The participant was asked to respond as quickly as possible to whether the central fish was facing to the left or right. Congruent trials were the ones with all five fish in the horizontal row pointing in the same direction and incongruent trials were the ones with the four distracting fishes pointing in the opposite direction of the central target fish. Reaction time of the congruent condition and of the incongruent condition were used to assess information processing speed, and the inhibition score (reaction time in incongruent conditions - reaction time in congruent conditions) was used as a measure of attentional control. Higher scores (reaction time) mean worse outcomes.
Flanker Visual Filtering Task (Christ, Kester, Bodner, & Miles, 2011) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The Flanker Visual Filtering Task was used to assess attentional control and information processing speed. Each trial showed a horizontal row of five fish. The participant was asked to respond as quickly as possible to whether the central fish was facing to the left or right. Congruent trials were the ones with all five fish in the horizontal row pointing in the same direction and incongruent trials were the ones with the four distracting fishes pointing in the opposite direction of the central target fish. Reaction time of the congruent condition and of the incongruent condition were used to assess information processing speed, and the inhibition score (reaction time in incongruent conditions - reaction time in congruent conditions) was used as a measure of attentional control. Higher scores (reaction time) mean worse outcomes.
Flanker Visual Filtering Task (Christ, Kester, Bodner, & Miles, 2011) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The Flanker Visual Filtering Task was used to assess attentional control and information processing speed. Each trial showed a horizontal row of five fish. The participant was asked to respond as quickly as possible to whether the central fish was facing to the left or right. Congruent trials were the ones with all five fish in the horizontal row pointing in the same direction and incongruent trials were the ones with the four distracting fishes pointing in the opposite direction of the central target fish. Reaction time of the congruent condition and of the incongruent condition were used to assess information processing speed, and the inhibition score (reaction time in incongruent conditions - reaction time in congruent conditions) was used as a measure of attentional control. Higher scores (reaction time) mean worse outcomes.
Reality Filtering Task (Liverani et al., 2017; Schnider, 2018) | Assessment at Time 1 (pre-intervention for "learning group"; pre-treatment as usual for "waiting group")
  The Reality Filtering task child-adapted version was used to assess recognition memory and orbitofrontal reality filtering. It consisted of a continuous recognition task composed of two runs with the same picture set but arranged in different order. Accuracy of the second run (D2) and Temporal Context Confusion index (TCC as defined by Schnider, 2018) measures reality filtering. Higher scores mean better outcomes.
Reality Filtering Task (Liverani et al., 2017; Schnider, 2018) | Assessment at Time 2 (immediately after the intervention for "learning group"; pre-intervention for "waiting group")
  The Reality Filtering task child-adapted version was used to assess recognition memory and orbitofrontal reality filtering. It consisted of a continuous recognition task composed of two runs with the same picture set but arranged in different order. Accuracy of the second run (D2) and Temporal Context Confusion index (TCC as defined by Schnider, 2018) measures reality filtering. Higher scores mean better outcomes.
Reality Filtering Task (Liverani et al., 2017; Schnider, 2018) | Assessment at Time 3 (3 months post-intervention for "learning group"; immediately after the intervention for "waiting group")
  The Reality Filtering task child-adapted version was used to assess recognition memory and orbitofrontal reality filtering. It consisted of a continuous recognition task composed of two runs with the same picture set but arranged in different order. Accuracy of the second run (D2) and Temporal Context Confusion index (TCC as defined by Schnider, 2018) measures reality filtering. Higher scores mean better outcomes.

SECONDARY OUTCOMES:
Neuroimaging acquisition | pre-intervention (Time 1 for "learning group"; Time 2 for "wainting group)
  (i) High resolution structural T1-weighted MP-RAGE (Magnetization Prepared Rapid Gradient Echo) sequence.
  (ii) Functional images were T2*-weighted with a multislice gradient-echo-planar imaging (EPI) sequence, including Resting-State fMRI data for which participants were asked to lie still with their eyes closed and engage into mind wandering and task-related activation paradigm (Flanker Visual Filtering Task, Reality Filtering task, Emotion Regulation task used to assessed emotional regulation functions (Samson, Kreibig, Soderstrom, Wade, & Gross, 2016) and the Recognition of Emotions in Contextual Scene task used to assessed facial emotional expression recognition based on contextual cues (Theurel et al., 2016)).
  (iii) Diffusion-weighted imaging (DWI) sequences were acquired with 1.3 mm3 isotropic voxels with four different shells.
Neuroimaging acquisition | immediately after the intervention (Time 2 for "learning group"; Time 3 for "wainting group)
  (i) High resolution structural T1-weighted MP-RAGE (Magnetization Prepared Rapid Gradient Echo) sequence.
  (ii) Functional images were T2*-weighted with a multislice gradient-echo-planar imaging (EPI) sequence, including Resting-State fMRI data for which participants were asked to lie still with their eyes closed and engage into mind wandering and task-related activation paradigm (Flanker Visual Filtering Task, Reality Filtering task, Emotion Regulation task used to assessed emotional regulation functions (Samson, Kreibig, Soderstrom, Wade, & Gross, 2016) and the Recognition of Emotions in Contextual Scene task used to assessed facial emotional expression recognition based on contextual cues (Theurel et al., 2016)).
  (iii) Diffusion-weighted imaging (DWI) sequences were acquired with 1.3 mm3 isotropic voxels with four different shells.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siffredi V, Liverani MC, Huppi PS, Freitas LGA, De Albuquerque J, Gimbert F, Merglen A, Meskaldji DE, Borradori Tolsa C, Ha-Vinh Leuchter R. The effect of a mindfulness-based intervention on executive, behavioural and socio-emotional competencies in very preterm young adolescents. Sci Rep. 2021 Oct 6;11(1):19876. doi: 10.1038/s41598-021-98608-2. PMID 34615893
- [Derived] Siffredi V, Liverani MC, Smith MM, Meskaldji DE, Stuckelberger-Grobety F, Freitas LGA, De Albuquerque J, Savigny E, Gimbert F, Huppi PS, Merglen A, Borradori Tolsa C, Leuchter RH. Improving executive, behavioural and socio-emotional competences in very preterm young adolescents through a mindfulness-based intervention: Study protocol and feasibility. Early Hum Dev. 2021 Oct;161:105435. doi: 10.1016/j.earlhumdev.2021.105435. Epub 2021 Jul 31. PMID 34507019